CLINICAL TRIAL: NCT01197677
Title: European Cardiovascular Magnetic Resonance Registry
Brief Title: European CMR Registry
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: Euro CMR
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Consecutive Patients Undergoing CMR
Keywords: CMR; Register; CAD; myocard scarring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. The main aim of the first specific protocol initiated by the European CMR registry, suspected CAD, is to demonstrate that patients presenting for work up of suspected coronary artery disease, which have a completely normal CMR scan will have a low risk for cardiovascular events.
2. The main aim of the second specific protocol initiated by the European CMR registry, HCM-SCD, will be to evaluate CMR for risk stratification in hypertrophic cardiomyopathy(HCM).
3. This registry is sought to collect data on the general use of CMR in the European clinical practice, its safety and its therapeutic implications in a high number of cases to 1) substantiate the clinical yield of CMR and 2) to define additional clinical questions worth to be investigated in detail as additional specific protocols in the future.

ELIGIBILITY:
Inclusion Criteria:

- European clinical practice: Consecutive patients with accomplished CMR.

-Suspected-CAD: Consecutive patients with suspected coronary artery disease undergoing a combined CMR protocol including evaluation of LV function, assessment of myocardial ische¬mia by adenosine stress perfusion or high-dose dobutamine CMR and detection of myocardial infarction using contrast-enhanced CMR.

- HCM-SCD: Consecutive patients with hypertrophic cardiomyopathy undergoing a combined CMR protocol including LV function, rest perfusion, and detection of myocardial scarring by contrast-enhanced CMR. The diagnosis of hypertrophic cardiomyopathy is based on the demonstration of a hypertrophied, non-dilated left ventricle (wall thickness of at least 15 mm in adults or the equivalent relative to body-surface area in children) in the absence of another cardiac or systemic disease capable of producing a similar degree of hypertrophy. In adult relatives of the patients with hypertrophic cardiomyo¬pathy, a wall thickness of 13 mm or more will be considered a criterion for diagnosis.

Exclusion Criteria:

* European clinical practice: None
* Suspected-CAD: Missing informed consent. Patients with known CAD by invasive coronary angiography or previous MI.
* HCM-SCD: Missing informed consent. Patients with known CAD by invasive coronary angiography or previous MI. Patients with left ventricular hypertrophy of other causes (e.g. hypertension, valvular heart disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing CMR (enrolled into the "European clinical practice"-part of the registry Consecutive patients with suspected coronary artery disease or with hypertrophic cardiomyopathy (enrolled into the specific protocols "suspected-CAD" or "HCM-SCD").
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
collect data from a large number of patients regarding the general use of CMR in European clinical practice, its safety and its therapeutic implications | 01/01/2009-

SECONDARY OUTCOMES:
to show that a normal CMR protocol (incl. LV wall motion at rest, stress ischemia, and scar detection) predicts a low risk of future cardiovascular events. | 01/01/2009
to evaluate if myocardial scarring assessed by contrast-enhanced CMR is a stronger predictor of adverse events during follow up than the general clinical markers of an adverse long term outcome in HCM. | 01/01/2009-

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Mahrholdt, MD, Principal Investigator — Robert-Bosch-Medical-Center, Stuttgart, Germany; Oliver Bruder, MD, Principal Investigator — Elisabeth-Hospital, Essen, Germany
Locations (10):
- Germany (7):
  - Klinikum Coburg, Coburg
  - Elisabeth Krankenhaus, Essen
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Krankenhaus Agatharied, Hausham
  - Klinikum Ludwigsburg-Bietigheim, Ludwigsburg
  - Robert Bosch Medical Centre, Stuttgart
  - Klinikum Traunstein, Traunstein
- Clinical Physiology Institute, Pisa, Italy
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Background] Bruder O, Wagner A, Mahrholdt H. Lessons Learned from the European Cardiovascular Magnetic Resonance (EuroCMR) Registry Pilot Phase. Curr Cardiovasc Imaging Rep. 2010 Jun;3(3):171-174. doi: 10.1007/s12410-010-9016-x. Epub 2010 Apr 13. PMID 20461126
- [Background] Wagner A, Bruder O, Schneider S, Nothnagel D, Buser P, Pons-Lado G, Dill T, Hombach V, Lombardi M, van Rossum AC, Schwitter J, Senges J, Sabin GV, Sechtem U, Mahrholdt H, Nagel E. Current variables, definitions and endpoints of the European cardiovascular magnetic resonance registry. J Cardiovasc Magn Reson. 2009 Nov 5;11(1):43. doi: 10.1186/1532-429X-11-43. PMID 19891768
- [Background] Bruder O, Schneider S, Nothnagel D, Dill T, Hombach V, Schulz-Menger J, Nagel E, Lombardi M, van Rossum AC, Wagner A, Schwitter J, Senges J, Sabin GV, Sechtem U, Mahrholdt H. EuroCMR (European Cardiovascular Magnetic Resonance) registry: results of the German pilot phase. J Am Coll Cardiol. 2009 Oct 6;54(15):1457-66. doi: 10.1016/j.jacc.2009.07.003. Epub 2009 Aug 13. PMID 19682818